CLINICAL TRIAL: NCT07152548
Title: Impact of Task-oriented Exercises and Mirror Therapy on Hand Functions Post Flexor Tendon Repair
Brief Title: Task-oriented Exercises and Mirror Therapy After Flexor Tendon Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Elshamy, Physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005415
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Flexor Tendon Injury
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Task-oriented exercises (Active Comparator)
  Interventions: Other: Task-oriented exercises
- Mirror Therapy (Active Comparator)
  Interventions: Other: Mirror Therapy
- Task-oriented exercises and mirror therapy (Active Comparator)
  Interventions: Other: Task-oriented exercises and mirror therapy

INTERVENTIONS:
Other: Task-oriented exercises and mirror therapy — Patients in this group will receive task-oriented exercises 3 sessions per week for 6 weeks.Therapy will include the following functional tasks: reaching, grasping or holding, lifting, placing objects, and counting fingers.Mirror therapy group: 3 sessions per week for 6 weeks.A mirror will be placed on the learning table, and exercises will be carried out by the patient looking into the mirror, where an unaffected limb would be placed in front of the mirror. Through looking into the mirror, the patient will assume the reflection of the unaffected limb is the affected limb. Exercises will be performed by hand opening and closing, wrist extension and flexion, squeezing, opposition, calculation, and finger flexion and extension.
  Arms: Task-oriented exercises and mirror therapy
Other: Task-oriented exercises — Patients in this group received task-oriented exercises 3 sessions per week for 6 weeks.Therapy included the following functional tasks: reaching, grasping or holding, lifting, placing objects, and counting fingers.
  Arms: Task-oriented exercises
Other: Mirror Therapy — Mirror therapy group 3sessions per week for 6 weeks. Mirror will be placed on the learning table and exercises will be carried out by the patient looking into the mirror where an unaffected limb would be placed in front of the mirror, through looking into the mirror patient will assume the reflection of the unaffected limb as the affected limb. Exercises will be performed hand opening and closing, wrist extension and flexion, squeezing, opposition, the calculation, finger flexion and extension.
  Arms: Mirror Therapy

SUMMARY:
The main objective of the study is to explore the effect of intervention with task-oriented exercises and mirror therapy on the outcomes of hand function post flexor tendon repair.

ELIGIBILITY:
Inclusion Criteria: - Ages of patients will range from 18 to 45 years. - All patients were working individuals before injury. - All patients will undergo zones of flexor tendon primary direct repair technique. - All patients will be referred by a surgeon before starting the study procedure. - All patients will enter the study having their informed consent. Exclusion Criteria: - Patients with associated vascular injuries requiring arterial repair. - Patients with associated soft tissue loss. - Patients with associated nerve injuries or bone fractures. - Patients with preexisting problems limiting joint motion. - Patients with tendon injuries in both hands. - Patients with diminished cognitive capacity. - Patients with a history of previously failed repair.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
ROM of wrist joints, proximal interphalangeal (PIP) joint and distal interphalangeal (DIP) joint of the involved digits of the involved hand for each patient. | pre- and post-6 weeks of treatment
  The standard values for AROM movements in the wrist and hand are: Wrist flexion: 80°-90° Wrist extension: 70°-90° Finger flexion: MCP: 85°-90° PIP: 100°-115° DIP: 80°-90° MCP extension: 30°-45°

SECONDARY OUTCOMES:
the Arabic version of the Michigan Hand Outcomes Questionnaire | pre- and post-6 weeks of treatment
  The Michigan Hand Outcomes Questionnaire (MHQ) is an example of a self-reporting outcome measure commonly used for the assessment of hand injuries. The MHQ was developed in 1998 and has become a very essential tool for the measurement of health status domains, activities of daily living, overall hand function, aesthetics, work performance, and satisfaction. The Michigan Hand Outcomes Measure comprises 37 items with rating scales ranging from 1 to 5.Every single domain is scored and converted to values that range from 0 to 100. A high score indicates better results, with the exception of pain, in which a high score indicates more intense pain. The total score was calculated as the sum of the six scores divided by six.

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Elshamy, B.Sc. of physical therapy, Principal Investigator — Cairo University
Locations (1):
- CairoU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Fernandez MV, Sarabia-Cobo CM, Sanchez-Labraca N. Cross-cultural adaptation, reliability, validity and responsiveness of the Michigan Hand Outcomes Questionnaire (MHQ-Sp) in Spain. J Orthop Surg Res. 2024 Apr 22;19(1):256. doi: 10.1186/s13018-024-04723-x. PMID 38649996
- [Background] Venkatramani H, Varadharajan V, Bhardwaj P, Vallurupalli A, Sabapathy SR. Flexor tendon injuries. J Clin Orthop Trauma. 2019 Sep-Oct;10(5):853-861. doi: 10.1016/j.jcot.2019.08.005. Epub 2019 Aug 19. PMID 31528057